CLINICAL TRIAL: NCT06057025
Title: Safety, Reactogenicity and Immunogenicity Study of the Drug "Sputnik Lite" for the Prevention of Coronavirus (COVID-19) Infection Caused by the SARS-CoV-2 Virus With Altered Antigenic Composition With Participation of Adult Volunteers.
Brief Title: Study of "Sputnik Lite" for the Prevention of COVID-19 With Altered Antigenic Composition.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gamaleya Research Institute of Epidemiology and Microbiology, Health Ministry of the Russian Federation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 14-Sputnik Lite / N-2023
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy patients (Experimental): Drug: Sputnik Light vector vaccine for the prevention of coronavirus infection caused by the SARS CoV-2 virus (with altered antigenic composition); A total of 50 people will be randomized and receive the study drug. A single intramuscular injection of the investigational medicinal product (IMP) will be performed.
  Interventions: Biological: "Sputnik Lite" vaccine for the prevention of COVID-19 with altered antigenic composition

INTERVENTIONS:
Biological: "Sputnik Lite" vaccine for the prevention of COVID-19 with altered antigenic composition — Single intramuscular injection of "Sputnik Lite" vaccine for the prevention of COVID-19 with altered antigenic composition.

SUMMARY:
Safety, reactogenicity and immunogenicity study of the drug "Sputnik Lite" for the prevention of coronavirus infection caused by the SARS-CoV-2 virus with altered antigenic composition with participation of adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

The study will include volunteers who meet all the specified criteria:

1. Subject's written informed consent to participate in the study;
2. Adult volunteer's men and women over 18 years old;
3. A negative test result for COVID-19, determined by PCR or express method before the introduction of the investigational medicinal product (IMP).
4. Consent to the use of effective methods of contraception during the entire period of participation in the study;
5. A negative pregnancy test based on the results of a urine test at a screening visit (for women with preserved reproductive potential);
6. Negative test for the presence of narcotic and psychostimulants in the urine at the screening visit;
7. Negative alcohol content test at the screening visit;
8. No contraindications to vaccination;
9. Absence of acute infectious and/or respiratory diseases for at least 14 days prior to inclusion in the study.

Exclusion Criteria:

Volunteers cannot be included in the study if there is at least one of the following criteria for non-inclusion:

1. No signed informed consent to participate in the study;
2. Therapy with steroids (with the exception of hormonal contraceptives and/or hormone replacement therapy) and / or immunoglobulins or other blood products that did not end 30 days before inclusion in the study;
3. Therapy with any immunosuppressive drugs completed less than 3 months before inclusion in the study;
4. Female subjects during pregnancy or lactation;
5. Acute coronary syndrome or stroke suffered less than one year before inclusion in the study;
6. Tuberculosis, chronic systemic infections according to anamnesis;
7. Burdened allergic anamnesis (the presence in the anamnesis of information about anaphylactic shock, Quincke's edema, polymorphic exudative eczema, serum sickness), hypersensitivity or allergic reactions to the administration of immunobiological drugs, known allergic reactions to the components of the drug, exacerbation of allergic diseases on the day of inclusion in the study;
8. The presence of neoplasms (ICD codes C00-D09) (according to the anamnesis);
9. Splenectomy (according to the anamnesis);
10. Neutropenia (decrease in the absolute number of neutrophils less than 1000/mm3), agranulocytosis, significant blood loss, severe anemia (hemoglobin less than 80 g/l), immunodeficiency - 6 months prior to inclusion in the study (according to the anamnesis);
11. Subjects with an active form of the disease caused by human immunodeficiency virus, syphilis, hepatitis B and C (according to anamnesis);
12. Anorexia, protein deficiency of any origin;
13. Alcoholism and drug addiction (according to anamnesis);
14. The subject's participation in any other interventional clinical trial (with the exception of rescreening in the current study) in the last 90 days;
15. Extensive tattoos at the injection sites (deltoid muscle area), which do not allow to assess the local reaction to the introduction of investigational medicinal product (IMP);
16. Any other condition of the subject of the study, which, in the opinion of the research doctor, may prevent the completion of the study in accordance with the protocol;
17. Vaccination against COVID-19 or transmitted coronavirus infection COVID-19 less than 6 months before screening;
18. Repeated administration of the Sputnik V vaccine, Sputnik Lite, or repeated administration of any other COVID-19 vaccine for more than three injections (Sputnik V vaccination plus Sputnik Lite revaccination);
19. Inability to read in Russian; inability or unwillingness to understand the essence of the study;
20. Any other conditions that limit the validity of obtaining informed consent or may affect the ability of the volunteer to participate in the study, affect the ability of the volunteer to participate in the study;
21. Staff of research centers (chief researcher and members of the research team) directly involved in the research and their family members.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of adverse events (AE) | Within 28 days after administration of the drug
  Occurrence of adverse events (AE)
Occurrence of serious adverse events (SAEs) | Throughout Study completion, until December 2024
  Occurrence of serious adverse events (SAEs)

IPD SHARING:
Plan to Share IPD: Undecided